CLINICAL TRIAL: NCT05488262
Title: Management in Intensive Care Unit of Life-threatening Keto-Acidosis
Acronym: MILKA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00455-38
Record Dates: First submitted 2022-07-25; First posted 2022-08-04 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Ketoacidosis
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients hospitalized in intensive care between January 2014 and December 2023 for ketoacidosis complicated by organ failure in participating departments.

DETAILED DESCRIPTION:
Analysis of patients with International Statistical Classification of Diseases and Related Health Problems coding compatible with inclusion

* Selection of patients eligible for inclusion based on review of medical records (verification of inclusion and non-inclusion criteria)
* Telephone contact and sending of the information letter on participation in the study and research of the patient's non-opposition to his participation and the processing of his data.
* Collection of retrospective data
* Phone call to collect prospective data

ELIGIBILITY:
Inclusion Criteria:

* Major (age ≥ 18 years old)
* Hospitalized in intensive care between January 2014 and December 2023 for ketoacidosis complicated by organ failure in the participating departments.
* Diagnosis of ketoacidosis judged to be the main cause of the severity of the clinical condition.
* Blood potential hydrogen < 7.15 and bicarbonates < 10mmol/L in the first 12 hours of treatment.
* Presenting at least one of the 3 organ failures during hospitalization among:
* Use of extra-renal purification for acute renal failure
* Administration of pressor amines
* Use of mechanical ventilation

Exclusion Criteria:

* Metabolic acidosis primarily of an origin other than ketonic
* Refusal to participate or opposition to the processing of their data
* Patient under guardianship or curators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care between January 2014 and December 2023 for ketoacidosis complicated by organ failure in participating departments.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
evaluate the incidence of mortality in intensive care units of patients hospitalized for severe diabetic ketoacidosis. | up to 6 months
  Percentage of mortality in intensive care units in patients admitted for ketoacidosis complicated by organ failure.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Avicenne, Bobigny
  - Louis Mourier, Colombes
  - Bicêtre, Le Kremlin-Bicêtre
  - Saint-Louis, Paris

IPD SHARING:
Plan to Share IPD: No